CLINICAL TRIAL: NCT03303001
Title: Subacromial Injection of High Volume Versus Conventional Steroid Injection Guided by Ultrasound in Shoulder Pain. Randomized Controlled Trial
Brief Title: Comparison Between Subacromial Infiltrations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Carlos A Acosta-Olivo, Professor, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OR17-00006
Record Dates: First submitted 2017-10-01; First posted 2017-10-05 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Subacromial Bursitis; Subacromial Impingement Syndrome; Rotator Cuff Impingement Syndrome
Keywords: subacromial infiltration; high volumen; shoulder pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Subacromial high volume infiltration (Experimental): This group received an subacromial infiltration guided by ultrasound, of 50 mL of solution. This solution mix: 2 mL of methylprednisolone (40 mg) plus 8 mL of lidocaine simple plus 10 mL of ropivacaine 7.5% plus 30 mL of saline solution.
  Interventions: Procedure: Subacromial high volume infiltration
- Subacromial conventional infiltration (Active Comparator): This group received an subacromial infiltration guided by ultrasound of 10 mL of solution. This solution mix: 2 mL of methylprednisolone (40 mg) plus 3 mL of lidocaine simple plus 5 mL of ropivacaine 7.5%
  Interventions: Procedure: Subacromial conventional infiltration

INTERVENTIONS:
Procedure: Subacromial high volume infiltration — This group will receive a high volume dose of a mix of methylprednisolone (40 mg in 2 mL) plus ropivacaine at 7.5% plus simple lidocaine plus saline solution for a total of 50 mL
  Other Names: subacromial infiltration
  Arms: Subacromial high volume infiltration
Procedure: Subacromial conventional infiltration — This group will receive a mix of solution of 2 mL of 40 mg of methylprednisolone plus 5 ml of ropivacaine at 7.5% plus 3 mL of lidocaine simple for a total of 10 ml
  Other Names: subacromial infiltration
  Arms: Subacromial conventional infiltration

SUMMARY:
The shoulder pain is commonly seeing in orthopedic consultation. Many patients was affected in activities of daily living and in laborer absent. One of the first treatment lines is the steroid infiltration for pain relieve, however in several times is only effective by a short period of time, and the symptoms usually appear again. One of the not known infiltration is the high volumen infiltration in subacromial space, this treatment appears to be an effective treatment for this patients.

DETAILED DESCRIPTION:
Shoulder pain is a common complaint in patients of all ages and activity levels, it is estimated that approximately 50% of the general population will experience at least one episode of shoulder pain over the course of a year. Shoulder pain has a general prevalence of 6.9-34%. The shoulder is the part of the upper extremity which is formed the proximal humerus, by the clavicle and the scapula, consisting in the shoulder griddle. The acromion is a bony process in the upper region of the scapula that articulates medially with the clavicle creating the acromioclavicular joint, at the same time forms the upper part of the shoulder joint. Between the humeral head and the acromion arch there is a space, the subacromial space, in which there are important structures for the proper functioning of the shoulder, among them, the subacromial bursa, the tendon of the rotator cuff and the tendon of the biceps brachii. The shoulder is the most mobile joint of all the body, therefore it is predisposed to suffer multiple injuries, including shoulder impingement syndrome, which has become one of the most frequent alterations of the musculoskeletal system. This pathology has an estimated prevalence of 43.7%. It is one of the most common causes of shoulder pain in the middle and advanced age patients.

Shoulder Impingement Syndrome is a condition in which structures in the subacromial space are chronically trapped between the humeral head and the acromion. It encompasses multiple conditions which includes partial rupture of the rotator cuff, rotator cuff tendinosis, calcified tendinitis or subacromial bursitis. All of these conditions may have a similar clinical picture and may be distinguishable by imaging of arthroscopy. The etiology of the syndrome is multifactorial, divided into extrinsic factors such as tendon overload, post trauma or repetitive microtraumas and intrinsic factors such as the vascularity of the tendon. There are also structural factors: anatomy of the acromion, subacromial osteophytes and acromioclavicular osteophytes; and functional factors: weakness of the rotator cuff, altered movement of scapula and ligament laxity increased. It is the result of a reduced space below the acromion. The most frequent clinical presentation will be insidious pain that can be installed in a period of days to months or after a trauma that can be irradiated to the side of the humerus. Usually the pain is nocturnal exacerbated by movements above the head or sleep on the affected shoulder and is attenuated by keeping the affected limb at rest.

Physical examination should assess muscular strength and ranges of motion. The general inspection should assess the presence of antalgic positions, muscular atrophy, asymmetries or sings of local inflammation. There is specific evidence for the evaluation of this pathology: Jobe's test, to evaluate de supraspinatus muscle, in which the patient is asked to perform 90° shoulder flexion, 30° abduction and external rotation and maintain the position against the shoulder resistance; Hawkins-Kennedy sign, for the subacromial impingement evaluation, with shoulder and elbow with 90° flexion perform rapid internal rotation of the shoulder, it is positive if it arouses with pain; Neer maneuver, for assessment of subacromial impingement, consists of the passive elevation of the extremity in abduction, flexion and internal rotation with stabilization of the scapula; Yocum´s maneuver, for assessment of subacromial impingement, the patient is asked to place the hand of the explored side in the contralateral shoulder and rises against resistance, it is positive if it causes pain. There are multiple differential diagnoses of this pathology, among which is adhesive capsulitis, cervical radiculopathy, glenohumeral instability, and acromioclavicular or glenohumeral osteoarthritis, among others.

The diagnosis is clinical and it is corroborated by imaging studies. Shoulder radiographs should be ordered in two positions to assess the morphology of the shoulder joint, to observe the distance between the humeral head to the acromion (11-14mm) and the evaluation of the acromioclavicular joint. Magnetic resonance imaging is the study of choice for evaluating shoulder impingement syndrome, where we will observe soft tissue structures that are part of the shoulder joint. Shoulder Impingement Syndrome is a pathology that causes pain and limitations to perform activities of daily living and evidence suggests that this condition is no self-limited, for this there are different alternatives of treatment. The aim of treatment is to decrease the pain and inflammation of soft tissues involved in the impingement in the subacromial space. Conservative treatment includes physical therapy, non-steroidal anti-inflammatory analgesics (NSAIDs) and subacromial infiltration. Surgical treatment includes shoulder arthroscopy to perform acromioplasty and thus release the subacromial space

Conservative Treatment

Physical Therapy Physical therapy is frequently implemented to reduce pain and improve shoulder function in this pathology. This must be carried out for at least six weeks. It includes cold-heat therapy, ultrasound, which has been shown to be of no benefit in the treatment of shoulder impingement and structural shoulder exercises, the aim of these treatment Is to reduce subacromial mechanical stress, to improve movement patterns and strengthening muscle fibers and thus prevent relapses, which have shown improvement in pain and function. Added to this it is recommended to avoid activities that are carried out above the head until the symptoms decrease.

Non-steroidal anti-inflammatory analgesics It is a frequent therapy in the treatment of this pathology. The effectiveness of NSAIDs in the treatment of shoulder impingement has not been demonstrated and potential complications have been observed with the use of long-term NSAIDs.

Shoulder Subacromial Injection It is a technique that consists of the direct application of an active principle in the subacromial space with the objective to suppress the inflammation and to diminish the pain. There are studies that show that there is a variation in the type and dose of steroids used in infiltration, in addition to that the number infiltrations also varied. Two studies conclude that there is an improvement in pain and range of motion with the use of this treatment.

Surgical Treatment Surgical treatment is indicated in patients who fail conservative treatment and continuous pain or in patients with complete rupture of the rotator cuff. Actually subacromial decompression with acromioplasty, osteophyte resection and bursectomy is performed by arthroscopy, in addition, to being able to observe the possible damage to the tendon of the rotator cuff, which, if present, can be repaired. It is currently mentioned that there is limited benefit with the conservative treatment established in the impingement syndrome, which is why new treatment options are being developed. A new treatment option is ultrasound-guided high-volume injection (HVIGI) in patients with shoulder impingement syndrome. Ultrasound-guided high-volume injection is a recent technique that involves injecting a high volume of fluid including a long-acting anesthetic and corticosteroids, guided by imaging (ultrasound). This technique has been used successfully and with good results in patellar tendinopathies, Achilles tendinopathies and subacromial impingement. High volume injection acts in different ways: breaks adhesions, stripping effect, stretch, has compression effect and also removes pain and promotes the healing of tendinopathy. Each injected component has different effect: the high volume breaks the adhesions, stretch and has drag effect; the long-acting anesthetic removes pain and the steroid prevents the formation of adhesions and promotes tendon healing

ELIGIBILITY:
Inclusion Criteria:

* Shoulder impingement syndrome
* Three months of history of pain and disability of the shoulder
* Failure to conservative initial treatment with NSAID's and rehabilitation

Exclusion Criteria:

* Rotator cuff tears
* Previous shoulder surgeries of any kind
* Glenohumeral or acromioclavicular arthritis
* Metabolic disease like diabetes mellitus or rheumatoid arthritis
* Previous infiltration in the past sixth months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Three months
  Measure the pain in patient, when 0 is no pain and 10 worst pain

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Three months
  Evaluates pain and function in 13 questions, with a scale from 0 to 10, normal shoulder is 0 and worst is 130
Simple Shoulder Test (SST) | Three months
  Twelve questions based on pain, function and range of motion, when 0 is an affected shoulder and 12 in a normal shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Acosta-Olivo, MD, PhD, Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Actually is an active study

REFERENCES:
- [Result] Morton S, Chan O, Ghozlan A, Price J, Perry J, Morrissey D. High volume image guided injections and structured rehabilitation in shoulder impingement syndrome: a retrospective study. Muscles Ligaments Tendons J. 2015 Oct 20;5(3):195-9. doi: 10.11138/mltj/2015.5.3.195. eCollection 2015 Jul-Sep. PMID 26605194
- [Result] Rossi F. Shoulder impingement syndromes. Eur J Radiol. 1998 May;27 Suppl 1:S42-8. doi: 10.1016/s0720-048x(98)00042-4. PMID 9652501
- [Result] Koester MC, George MS, Kuhn JE. Shoulder impingement syndrome. Am J Med. 2005 May;118(5):452-5. doi: 10.1016/j.amjmed.2005.01.040. PMID 15866244
- [Result] Chard MD, Sattelle LM, Hazleman BL. The long-term outcome of rotator cuff tendinitis--a review study. Br J Rheumatol. 1988 Oct;27(5):385-9. doi: 10.1093/rheumatology/27.5.385. PMID 3179628
- [Result] Green S, Buchbinder R, Hetrick S. Physiotherapy interventions for shoulder pain. Cochrane Database Syst Rev. 2003;2003(2):CD004258. doi: 10.1002/14651858.CD004258. PMID 12804509
- [Result] Buchbinder R, Green S, Youd JM. Corticosteroid injections for shoulder pain. Cochrane Database Syst Rev. 2003;2003(1):CD004016. doi: 10.1002/14651858.CD004016. PMID 12535501
- [Result] Petri M, Dobrow R, Neiman R, Whiting-O'Keefe Q, Seaman WE. Randomized, double-blind, placebo-controlled study of the treatment of the painful shoulder. Arthritis Rheum. 1987 Sep;30(9):1040-5. doi: 10.1002/art.1780300911. PMID 3311051
- [Result] Wheeler PC, Mahadevan D, Bhatt R, Bhatia M. A Comparison of Two Different High-Volume Image-Guided Injection Procedures for Patients With Chronic Noninsertional Achilles Tendinopathy: A Pragmatic Retrospective Cohort Study. J Foot Ankle Surg. 2016 Sep-Oct;55(5):976-9. doi: 10.1053/j.jfas.2016.04.017. Epub 2016 Jun 7. PMID 27286927